CLINICAL TRIAL: NCT02945241
Title: Impact of Cystatin-C C-guided Vancomycin Dosing Recommendation on Target Trough Achievement and Clinical Outcomes in Critically Ill Adults
Brief Title: Cystatin-C C-guided Vancomycin Dosing in Critically Ill Patients: A Quality Improvement Project
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erin Barreto, Assistant Professor of Pharmacy and Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-002808
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Methicillin-resistant Staphylococcus Aureus; Sepsis; Critical Illness
MeSH Terms: conditions — Sepsis; Critical Illness | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystatin C-guided vancomycin dosing algorithm (Experimental): Cystatin C is an endogenous cysteine proteinase inhibitor produced by all nucleated cells and a biomarker used routinely to estimate glomerular filtration rate either alone or in combination with creatinine. This new dosing algorithm includes patient weight, individualized goal trough concentration, and glomerular filtration rate (expressed with the CKD-EPI creatinine-cystatin C equation in mL/min) to determine dose and frequency.
  Interventions: Drug: Vancomycin; Other: Cystatin C dosing algorithm
- Creatinine clearance guided vancomycin dosing (Other): Historical controls for the quality improvement project had doses based on weight and interval established with the creatinine clearance using the Cockcroft-Gault equation.
  Interventions: Drug: Vancomycin; Other: Creatine clearance dosing algorithm

INTERVENTIONS:
Drug: Vancomycin — Intravenous
  Other Names: Vancocin
Other: Cystatin C dosing algorithm — Expressed in milliliters per minute
  Arms: Cystatin C-guided vancomycin dosing algorithm
Other: Creatine clearance dosing algorithm — Vancomycin dosing algorithm based on creatinine clearance, expressed in milliliters per minute
  Other Names: Cockcroft-Gault
  Arms: Creatinine clearance guided vancomycin dosing

SUMMARY:
Determine if a cystatin C-inclusive vancomycin dosing algorithm improved target trough achievement compared to creatinine clearance-guided vancomycin therapy in critically ill patients.

DETAILED DESCRIPTION:
This is a prospective, quality improvement study that evaluated critically ill patients initiated on intravenous vancomycin. Between January 2012 through October 2013, vancomycin was dosed at 15-20mg/kg at an interval guided by creatinine clearance using the Cockcroft Gault equation (control arm). Steady state trough concentrations were assessed prior to the 4th dose of a consistent regimen and compared to the individualized target trough range (10-15mg/L or 15-20mg/L) appropriate for the suspected or documented source of infection. Given low overall trough achievement observed with standard care, a quality improvement project was undertaken. After approval by local clinical practice committees with representation from the Division of Infectious Diseases, Pharmacy and Critical Care, a quality improvement project was undertaken to implement a new vancomycin dosing nomogram with dosing intervals based on the Chronic Kidney Disease Epidemiology Collaborative (CKD-EPI) creatinine-cystatin GFR equation, expressed in mL/min. After structured education was provided, the dosing algorithm was rolled out from December 2013 through May 2015 (intervention arm). Steady state target vancomycin trough achievement was compared between study arms with and without adjustment for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in one of three intensive care units at Mayo Clinic in Rochester, Minnesota
* Suspected or documented gram-positive infection
* Prescribed IV vancomycin at a consistent dose and scheduled with 8, 12, or 24 hour Vancomycin dosing interval

Exclusion Criteria:

* Vulnerable population
* Received greater than 1 dose of Vancomycin in the 96 hours before ICU admission
* Baseline glomerular filtration rate (GFR) of less than 20 milliliters/minute
* Undergoing renal replacement therapy
* Body mass index > 40kg/m2
* Weight < 40kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Vancomycin target trough achievement | Baseline
  The percentage of initial steady state troughs within the target range.

SECONDARY OUTCOMES:
Length of stay (hospital and ICU) | Baseline
Acute kidney injury (AKI) and renal replacement therapy | 7-days
  New onset AKI, defined as KDIGO stage II or greater AKI, within 48-hours of and within 7-days of vancomycin initiation
Treatment failure | 7-days
  Treatment failure in patients with confirmed gram-positive infection after at least 48-hours of vancomycin therapy and within 7-days
Infection recurrence | 28-days
  New onset of infection within 28-days among patients with confirmed gram-positive infection

CONTACTS AND LOCATIONS:
Overall Officials: Erin Frazee, PharmD, RPh, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frazee EN, Rule AD, Herrmann SM, Kashani KB, Leung N, Virk A, Voskoboev N, Lieske JC. Serum cystatin C predicts vancomycin trough levels better than serum creatinine in hospitalized patients: a cohort study. Crit Care. 2014 May 29;18(3):R110. doi: 10.1186/cc13899. PMID 24887089